CLINICAL TRIAL: NCT06826443
Title: A Comparative Evaluation of Mosapride Versus Metoclopramide for Enteral Feeding Intolerance in Critically Ill Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Mohamed El Mokadem, Lecturer of Pharmacy Practice and Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM000185
Record Dates: First submitted 2025-02-06; First posted 2025-02-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Enteral Feeding Intolerance
MeSH Terms: interventions — mosapride; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mosapride citrate group (Active Comparator): These patients will receive Mosapride citrate (5 mg) three times daily for 7 days.
  Interventions: Drug: Mosapride Citrate Tablets
- Metoclopramide (Active Comparator): These patients will receive metoclopramide (10 mg) three times daily for 7 days.
  Interventions: Drug: Metoclopramide 10mg

INTERVENTIONS:
Drug: Mosapride Citrate Tablets — Prokinetic Drug
  Arms: Mosapride citrate group
Drug: Metoclopramide 10mg — Prokinetic Drug
  Arms: Metoclopramide

SUMMARY:
Caring for critically ill patients in an intensive care unit (ICU) is considered a standard of care. According to the Society of Critical Care Medicine (SCCM), as a function of the complex nature of the care provided in the ICU, the ideal method to provide support to the critically ill involves the participation of a multi-professional staff.

Provision of nutrition support to the critically ill is now established as an essential part of patient care where aiming toward 100% of the predicted target may have resulted in reduced mortality and increased ventilator-free days in those who are premorbid malnourished. Despite these reported benefits, clinicians continue to deliver little more than half of the enteral nutrition (EN) they plan to provide, due to gastric motility disorders, patient intolerance and clinical interruptions. Also despite the availability of numerous clinical practice guidelines (CPGs) focused on feeding critically ill patients, observational studies have consistently demonstrated persistent and significant gaps between guideline recommendations and actual nutrition practice. Consequently, underfeeding is prevalent in the intensive care unit (ICU), with patients on average receiving only 60 % of the calories that are prescribed. Moreover, Among the barriers to adequate nutritional supply in the ICU which contributes to nutritional status deterioration, gastrointestinal disorders causing enteral feed intolerance are the most important and the most often mentioned in the literature. when gastric emptying was measured in critically ill patients, 46 % of them had evidence of delayed gastric emptying. Untreated slow gastric emptying has a plethora of clinical consequences such as vomiting, aspiration of gastric contents, pneumonia, and contributes significantly to the frequent interruptions and cessation of EN in the ICU, which results in inadequate nutritional delivery. Studies have shown an association between feeding intolerance, prolonged intensive care unit (ICU) stay, and increased risk of death.

Guidelines for the provision and assessment of nutrition support therapy in the adult critically ill patients has demonstrated the importance of the use of prokinetic drugs to improve tolerance to gastric feeding in critically ill patients and achieve earlier discharge.

Prokinetic drugs act by promoting gastric motility, increase gastric emptying, prevent the retention and reflux of gastric contents and thus provide symptomatic relief.

Most of the prokinetic drugs are efficacious with prokinetic activity but the matter of major concern is their side effect profile. The most commonly used agent is metoclopramide. Although it is the most commonly used prokinetic to treat delayed gastric emptying and facilitate early enteral feeding, adverse complications limit its use including tachyphylaxis, tardive dyskinesia on long term use and QT prolongation predisposing to cardiac arrhythmias. Several drug targets have been identified to develop new promotility agents and several new medications are under investigation to overcome the side effects caused by most of the prokinetics .

Mosapride is another available prokinetic agent that enhances gastric motility through serotonin receptor agonism; resulting in prokinetic effects. It accelerates gastric emptying, improves gastric tension and sensitivity, and has anti-emetic action.

The aim of the current study is to compare the effectiveness as well as the safety of Mosapride against metoclopramide as the first line treatment for feeding intolerance in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging between 18 and 60 years (of both sexes)
* Patients admitted to the ICU and are expected to stay in the ICU for not less than 7 days
* Patients prescribed enteral feeding.

Exclusion Criteria:

The following patients are

* Age less than 18 years or more than 60 years.
* Patients who had previous upper gastrointestinal tract surgery, obstruction, hemorrhage or history of GI disease.
* Patients who are clinically significant hepatic dysfunction. (>3 times above the upper end of normal range of bilirubin, γ-glutamyl transferase, aspartate transaminase, or lactate dehydrogenase)
* Patients who are on regular use of H2 blockers, prokinetic, proton pump inhibitor or anticholinergic agents for previous 4 weeks.
* Patients with arrhythmia or atrioventricular blocks.
* Patients with any condition or comorbid disease that might interfere with gastric emptying such as diabetes.
* Patients with head injuries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Gastric residual volume will be measured by ultrasonography | GRV will be measured daily for the duration of therapy which is 7 days
  the gastric residual volume will be assessed by ultrasonography on daily basis for the duration of the study period

SECONDARY OUTCOMES:
Incidence of infectious complications such as pneumonia or any other infection complication will be assessed throughout the study period | Incidence of infectious complications will be assessed for the 7 days study period
Length of intensive care unit (ICU) stay will be assessed from the day of admission to ICU till the day of discharge from ICU | Length of ICU stay will be assessed from the day of admission to the ICU till the day of discharge from ICU
Any Adverse drug event as abdominal pain, QT prolongation and cardiac side effects that occur within the study period will be recorded throughout the study period | adverse drug events will be recorded for the study period of 7 days
Determining the adequacy of enteral nutrition will be assessed by measuring the enteral nutrition volume ratio at base line and at the end of the study period | Determining the adequacy of enteral nutrition will be assessed on daily base for the duration of study period of 7 days
  the adequacy of enteral nutrition will be assessed by measuring the enteral nutrition volume ratio (the ratio of the actual received to the prescribed enteral nutrition volume ) at baseline of the study and at the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Matarya Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charoensareerat T, Bhurayanontachai R, Sitaruno S, Navasakulpong A, Boonpeng A, Lerkiatbundit S, Pattharachayakul S. Efficacy and Safety of Enteral Erythromycin Estolate in Combination With Intravenous Metoclopramide vs Intravenous Metoclopramide Monotherapy in Mechanically Ventilated Patients With Enteral Feeding Intolerance: A Randomized, Double-Blind, Controlled Pilot Study. JPEN J Parenter Enteral Nutr. 2021 Aug;45(6):1309-1318. doi: 10.1002/jpen.2013. Epub 2020 Oct 2. PMID 32895971